CLINICAL TRIAL: NCT01199432
Title: A Phase Ⅳ Randomized Clinical Trial of Comparative Efficiency of Three Regimen, CEFci, CEF and EC as Neoadjuvant Chemotherapy for Primary Breast Cancer
Brief Title: Comparative Efficiency of Three Regimen, CEFci, CEF and EC as Neoadjuvant Chemotherapy for Primary Breast Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tao OUYANG (Other)
Responsible Party: Sponsor-Investigator, Tao OUYANG, Chairman of Breast Center, Peking University
Organization: Peking University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCP06
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Breast Cancer
Keywords: Primary Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — EC regimen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group B(CEF) (Experimental)
  Interventions: Drug: 5-FU（intravenous bolus）+epirubicin+cyclophosphamide
- Group A(CEFci) (Experimental)
  Interventions: Drug: 5-FU（intravenous infusion）+epirubicin+cyclophosphamide
- Group C(EC) (Active Comparator)
  Interventions: Drug: epirubicin+cyclophosphamide

INTERVENTIONS:
Drug: 5-FU（intravenous infusion）+epirubicin+cyclophosphamide — 5-FU 200mg/m2 per day from day 1 to day 28 （Continuous intravenous infusion）; epirubicin 65mg/m2 per day on day 1 and day 8 and cyclophosphamide 500mg/m2 per day on day 1 and day 8 ; every 28 days as a cycle. Total four cycles is needed
  Other Names: CEFci
  Arms: Group A(CEFci)
Drug: 5-FU（intravenous bolus）+epirubicin+cyclophosphamide — 5-FU 500mg/m2 per day on day 1 and day 8（intravenous bolus）; epirubicin 65mg /m2 per day on day 1 and day 8 and cyclophosphamide 500mg/m2 per day on day 1 and day 8 ; every 28 days as a cycle. Total four cycles is needed.
  Other Names: CEF
  Arms: Group B(CEF)
Drug: epirubicin+cyclophosphamide — epirubicin 65mg/m2 per day on day 1 and day 8 and cyclophosphamide 500mg/m2 per day on day 1 and day 8 ; every 28 days as a cycle. Total four cycles is needed.
  Other Names: EC
  Arms: Group C(EC)

SUMMARY:
This is a phase IV, prospective, single-center, open-label, randomized, controlled study. Eligible patients are randomly assigned into three groups. The investigators propose to evaluate and compare the efficacy and safety of different neoadjuvant chemotherapies in women with primary breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, age ≦ 65 years old
* Histologically or cytologically confirmed primary breast cancer by core biopsy
* Disease stage appropriate for neoadjuvant chemotherapy (T2～T3，N0～2，M0)
* No previous treatment for breast cancer
* No history of other malignancies
* No currently uncontrolled diseased (e.g., ongoing cardiac dysrhythmias, unstable diabetes) or active infection
* No history of other malignancies
* No currently uncontrolled diseased or active infection
* Not pregnant or breast feeding, and on appropriate birth control if of child-bearing potential
* Adequate cardiovascular function reserve without a myocardial infarction within the past six month
* Adequate hematologic function with:

  1. Absolute neutrophil count (ANC) ≥ 1500/mm3
  2. Platelets ≥ 100,000/ mm3
  3. Hemoglobin ≥ 10 g/dL
* Adequate hepatic and renal function with:

  1. Serum bilirubin ≤ 1.5×UNL
  2. Alkaline phosphatase and alanine aminotransferase (ALT) ≤ 2.5 x ULN.
  3. Serum creatinine ≤ 1.7 mg/dl
* Knowledge of the investigational nature of the study and Ability to give informed consent
* Ability and willingness to comply with study procedures

Exclusion Criteria:

* Known or suspected distant metastases
* Concurrent malignancy or history of other malignancy
* Uncontrolled diseases or active infection
* Hepatic or renal dysfunction as detailed above
* Geographical, social, or psychological problems that would compromise study compliance
* Known or suspected hypersensitivity to cyclophosphamide, epirubicin and fluorouracil

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Estimated)
Dates: Start 2010-10; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pathologic complete response （PCR） | up to four weeks after surgery
  pathological evaluation by Miller & Payne Grading System. Pathological complete response (pCR) was defined as no histological evidence of invasive tumor cells in the breast. The presence of DCIS alone was considered as pCR (G5). Residual cancer consisting of scattered tumor cells, not directly measurable, was reported as near pCR (G4)

SECONDARY OUTCOMES:
Number of Participants with Ⅲ° and Ⅳ° Adverse Events According to NCI-CTC | at the last day of every chemotherapy cycle
  All adverse events that occur after the initiation of the treatment will be handled with utmost attention, and carefully documented. Investigator will identify the adverse events according to National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 3.0, the Common Terminology Criteria for Adverse Events.Development of a severe side effect will be an indication for drop-outs.
Number of patients undergoing breast conserving surgery | up to a week after operation

CONTACTS AND LOCATIONS:
Overall Officials: Tao Ouyang, Doctor, Study Chair — Beijing Cancer Hospital Breast Center
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China